CLINICAL TRIAL: NCT00087126
Title: A Phase II Evaluation of Weekly Topotecan Hydrochloride (Hycamtin®, NSC #609699) in the Treatment of Persistent or Recurrent Carcinoma of the Cervix
Brief Title: Topotecan in Treating Women With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0127U; GOG-0127U; CDR0000372930 (Other: CDR)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2015-05

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topotecan (Experimental): Topotecan weekly
  Interventions: Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well topotecan works in treating women with persistent or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of topotecan in patients with persistent or recurrent carcinoma of the cervix that failed higher priority treatment protocols.
* Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive topotecan IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patient are followed for every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the cervix

  * Squamous cell or nonsquamous cell
  * Persistent or recurrent disease
  * Documented disease progression
* Measurable disease

  * At least 1 unidimensionally measurable target lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
  * Tumors within a previously irradiated field are considered non-target lesions unless disease progression is documented or a biopsy is obtained to confirm persistent disease at least 90 days after completion of prior radiotherapy
* Must have received 1 prior systemic chemotherapy regimen for persistent or recurrent squamous cell or nonsquamous cell carcinoma of the cervix

  * Chemotherapy administered with primary radiotherapy as a radiosensitizer is not considered a systemic chemotherapy regimen
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Other

* Sensory or motor neuropathy ≤ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* One prior non-cytotoxic (biologic or cytostatic) regimen for recurrent or persistent disease allowed, including, but not limited to, the following:

  * Monoclonal antibodies
  * Cytokines
  * Small-molecule inhibitors of signal transduction
* At least 3 weeks since prior biologic or immunologic agents for cervical cancer
* No concurrent prophylactic growth factors, including filgrastim (G-CSF), sargramostim (GM-CSF), or pegfilgrastim
* No concurrent prophylactic thrombopoietic agents

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen (either with single or combination cytotoxic drug therapy)
* No prior topotecan

Endocrine therapy

* At least 1 week since prior hormonal therapy for cervical cancer
* Concurrent hormone replacement therapy allowed

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* Recovered from prior surgery

Other

* At least 3 weeks since other prior therapy for cervical cancer
* No prior cancer therapy that would preclude study participation

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-02; Primary Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James V. Fiorica, MD, Study Chair — Sarasota Memorial Hospital
Locations (27):
- United States (27):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Olive View - UCLA Medical Center Foundation, Sylmar, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island

REFERENCES:
- [Result] Fiorica JV, Blessing JA, Puneky LV, Secord AA, Hoffman JS, Yamada SD, Buekers TE, Bell J, Schilder JM; Gynecologic Oncology Group. A Phase II evaluation of weekly topotecan as a single agent second line therapy in persistent or recurrent carcinoma of the cervix: a Gynecologic Oncology Group study. Gynecol Oncol. 2009 Nov;115(2):285-9. doi: 10.1016/j.ygyno.2009.07.024. Epub 2009 Sep 2. PMID 19726073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on January 3, 2005 and was closed to accrual on October 29, 2007.
Groups:
- Topotecan Hydrochloride: Topotecan hydrochloride 3.0 mg/m² IV over 30 minutes every 7 days for 21 days; 7 days off (cycle = 28 days)
Period: Overall Study
Arm/Group | Topotecan Hydrochloride
Started | 27
Completed (Eligible and treated patients) | 25
Not Completed | 2
Not completed — Ineligible - second primary | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 25
Age, Customized [Number; unit: participants]
  <40 years | 4
  40-49 years | 10
  50-59 years | 8
  60-69 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; every 6 months thereafter until disease progression for up to 5 years.
Population: Eligible and treated patients with sufficient follow-up assessments to evaluate response
Measure: Number; unit: participants
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 22
participants
  Partial response | 0
  Complete response | 0

2. Primary Outcome: Number of Participants With Adverse Effects as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: All participants assessed by CTCAE v3 (Common Terminology Criteria for Adverse Events version 3.0) including grade 0 (the number of participants not affected by the Adverse Event).
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Population: Eligible and treated patients
Measure: Number; unit: participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25
participants
  Leukopenia | 6 | 4 | 9 | 5 | 1
  Thrombocytopenia | 16 | 4 | 3 | 0 | 2
  Neutropenia | 9 | 8 | 4 | 2 | 2
  Transfusions | 24 | 0 | 0 | 1 | 0
  Anemia | 1 | 4 | 12 | 7 | 1
  Hemorrhage | 24 | 1 | 0 | 0 | 0
  Nausea/Vomiting | 13 | 7 | 4 | 1 | 0
  Other gastrointestinal | 12 | 4 | 6 | 3 | 0
  Genito urinary | 22 | 2 | 1 | 0 | 0
  Neurotoxicity | 19 | 3 | 2 | 0 | 1
  Pain | 19 | 4 | 1 | 0 | 1
  Pulmonary | 24 | 0 | 0 | 1 | 0
  Infection | 22 | 0 | 0 | 3 | 0
  Constitutional | 8 | 5 | 7 | 3 | 2
  Metabolic | 22 | 2 | 1 | 0 | 0
  Dermatologic | 22 | 3 | 0 | 0 | 0
  Alopecia | 17 | 7 | 1 | 0 | 0
  Renal | 21 | 3 | 1 | 0 | 0
  Alkaline Phosphatase | 23 | 2 | 0 | 0 | 0
  Vascular | 24 | 0 | 0 | 1 | 0
  Lymphatics | 24 | 0 | 0 | 1 | 0
  Lymphopenia | 24 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | Topotecan Hydrochloride
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan Hydrochloride (N=25)
Fatigue (General disorders) | 1
Death No Ctcae Term - Death Nos (Not Otherwise Specified) (General disorders) | 1
Infection with Normal Or Grade 1 Or 2 Absolute Neutrophil Count: Lung (Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Central nervous system ischemia (Nervous system disorders) | 1
Diplopia (Eye disorders) | 1
Pain: Extremity-Limb (General disorders) | 1
Pain: Back (General disorders) | 1
Stricture, Anastomotic, Genitourinary - Ureter (Renal and urinary disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topotecan Hydrochloride (N=25)
Leukopenia (Blood and lymphatic system disorders) | 19
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 16
Transfusions (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 24
Hemorrhage (Vascular disorders) | 1
Nausea/Vomiting (Gastrointestinal disorders) | 12
Other gastrointestinal (Gastrointestinal disorders) | 13
Genito urinary (Renal and urinary disorders) | 3
Neurotoxicity (Nervous system disorders) | 6
Pain (General disorders) | 6
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 3
Constitutional (General disorders) | 17
Metabolic (Metabolism and nutrition disorders) | 3
Dermatologic (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 8
Renal (Renal and urinary disorders) | 4
Alkaline phosphatase (Investigations) | 2
Vascular (Vascular disorders) | 1
Lymphatics (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less